CLINICAL TRIAL: NCT02212236
Title: Development and Evaluation of a Psychological Intervention to Alleviate Distress During Haematopoietic Stem-cell Transplantation
Brief Title: Psychological Intervention for Distress During HSCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Nottingham University Hospitals NHS Trust (Other); Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 14069
Record Dates: First submitted 2014-08-04; First posted 2014-08-08 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Psychological Distress; Haematopoietic Stem Cell Transplantation; Bone Marrow Transplantation
Keywords: Distress; Depression; Anxiety; Stress; Coping; Illness perceptions; Stem cell transplantation; Bone marrow transplantation
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psychological preparation + TAU (Experimental): TAU=treatment as usual
  Interventions: Other: Psychological preparation
- Treatment as usual (No Intervention): Usual care including medication, nursing, and psychologist support.

INTERVENTIONS:
Other: Psychological preparation — Ninety-minute, group-based psychological preparation delivered prior to haematopoietic stem cell transplantation aiming at alleviating psychological distress during the procedure by enhancing perceptions of the procedure and fostering more helpful coping.
  Arms: Psychological preparation + TAU

SUMMARY:
This Phase II trial aims to evaluate a new psychological intervention to alleviate distress during haematopoietic stem cell transplantation (HSCT) together with examining feasibility.

HSCT is a complex procedure aimed at a range of haematological and autoimmune illnesses. Over 3,000 individuals undergo the procedure every year in the UK with substantial benefits. However, it is very costly, intensive, and has a range of debilitating side effects. Consequently, patients often experience considerable distress, which can impede recovery.

A 90-minute, group-based intervention has been developed to address this need based on psychological theory of adjustment to illness-related difficulties. It is delivered by the transplant team and involves provision of information to foster more helpful perceptions about HSCT and facilitating more helpful coping with its difficulties. To evaluate the effectiveness of the intervention in alleviating distress, 60 patients about to undergo HSCT at two sites (Sheffield & Nottingham) will be randomly allocated into two groups. Patients in the intervention group will receive the new intervention prior to transplantation together with treatment as usual (TAU) while patients in the control group will receive TAU alone. Participants and the researcher collecting the data will be blind to the allocation.

Demographic and relevant clinical information will be recorded at the end of participation to ensure effectiveness of randomisation. For both groups, resilience, distress, coping, and procedure-related perceptions will be measured at four time points: (i) prior to the intervention/transplantation, (ii) day of transplant, (iii) two weeks following the transplant, and (iv) four weeks following the transplant. It is hypothesised that patients in the intervention group will experience higher resilience and lower distress compared to controls and that this difference will be mediated by procedure-related perceptions and coping. A subgroup of participants of those randomised to the group intervention will be invited to participate in a feedback interview at the end.

ELIGIBILITY:
Inclusion Criteria:

* patients referred for HSCT as treatment for haematological malignancy
* age of 18 years or older
* sufficient command of the English language or access to suitable support to comprehend materials and participate in the group and data collection over the telephone
* informed consent
* permission will also be sought by the patient's Consultant Haematologist once clients have consented

Exclusion Criteria:

* Consent withdrawn
* Consultant Haematologist raises concern regarding participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Depression Anxiety Stress Scales (DASS-21) | Baseline
  Assesses presence of depression, anxiety, stress, and overall distress; 21 items, Likert-type.
Depression Anxiety Stress Scales (DASS-21) | Day 0 (transplant day)
  Assesses presence of depression, anxiety, stress, and overall distress; 21 items, Likert-type.
Depression Anxiety Stress Scales (DASS-21) | Day 14
  Assesses presence of depression, anxiety, stress, and overall distress; 21 items, Likert-type.
Depression Anxiety Stress Scales (DASS-21) | Day 28
  Assesses presence of depression, anxiety, stress, and overall distress; 21 items, Likert-type.

SECONDARY OUTCOMES:
Brief Resilience Scale (BRS) | Baseline
  Assesses resilience; 6 items, Likert-type.
Brief Resilience Scale (BRS) | Day 0 (transplant day)
  Assesses resilience; 6 items, Likert-type.
Brief Resilience Scale (BRS) | Day 14
  Assesses resilience; 6 items, Likert-type.
Brief Resilience Scale (BRS) | Day 28
  Assesses resilience; 6 items, Likert-type.
Brief Coping with Problems Experienced scale (COPE) | Baseline
  Assesses coping styles; 28-item, Likert-type.
Brief Coping with Problems Experienced scale (COPE) | Day 0 (transplant day)
  Assesses coping styles; 28-item, Likert-type.
Brief Coping with Problems Experienced scale (COPE) | Day 14
  Assesses coping styles; 28-item, Likert-type.
Brief Coping with Problems Experienced scale (COPE) | Day 28
  Assesses coping styles; 28-item, Likert-type.
Brief Illness Perceptions Questionnaire (IPQ) | Baseline
  Assesses illness perceptions, adapted for haematopoietic stem cell transplantation; 9-item, Likert-type.
Brief Illness Perceptions Questionnaire (IPQ) | Day 0 (transplant day)
  Assesses illness perceptions, adapted for haematopoietic stem cell transplantation; 9-item, Likert-type.
Brief Illness Perceptions Questionnaire (IPQ) | Day 14
  Assesses illness perceptions, adapted for haematopoietic stem cell transplantation; 9-item, Likert-type.
Brief Illness Perceptions Questionnaire (IPQ) | Day 28
  Assesses illness perceptions, adapted for haematopoietic stem cell transplantation; 9-item, Likert-type.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Schröder, PhD, Principal Investigator — University of Nottingham
Locations (2):
- United Kingdom (2):
  - Nottingham City Hospital, Nottingham, Nottinghamshire
  - Royal Hallamshire Hospital, Sheffield, South Yorkshire